CLINICAL TRIAL: NCT04127708
Title: Akasaray University
Brief Title: Tinnitus and Acupuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, ihsan kuzucu, ent, Aksaray University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tinnitusacupuncture
Record Dates: First submitted 2019-09-21; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Tinnitus, Subjective
Keywords: tinnitus; acupuncture; otology; prospective study
MeSH Terms: conditions — Tinnitus | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham acupuncture (Placebo Comparator): Ten acupuncture sessions were applied over five weeks. In this study, acupuncture style is the traditional Chinese model, acupuncture was performed on 11 acupuncture points (TE21, SI19, GB2, TE22, ST7, TE17, GB20 of the affected side, and GB20, TE05, KI3 of both sides) using sterile, single-use, 0.25 mm thick, 40 mm long needles (Dongbang Medical Co., Boryeong, Korea). The acupuncture points were selected by taking previous studies as reference. The depth of the needle differed depending on the anatomical structure of the participant and the nature of the acupuncture points, but it was approximately 5-10 mm. The acupuncture needles were applied until the participant experienced de-qi and removed after 20 minutes.
  Interventions: Biological: acupuncture
- acupuncture (Active Comparator): en acupuncture sessions were applied over five weeks. In this study, acupuncture style is the traditional Chinese model, acupuncture was performed on 11 acupuncture points (TE21, SI19, GB2, TE22, ST7, TE17, GB20 of the affected side, and GB20, TE05, KI3 of both sides) using sterile, single-use, 0.25 mm thick, 40 mm long needles (Dongbang Medical Co., Boryeong, Korea). The acupuncture points were selected by taking previous studies as reference. The depth of the needle differed depending on the anatomical structure of the participant and the nature of the acupuncture points, but it was approximately 5-10 mm. The acupuncture needles were applied until the participant experienced de-qi and removed after 20 minutes.
  Interventions: Biological: acupuncture

INTERVENTIONS:
Biological: acupuncture — acupuncture group and control group
  Other Names: sham group

SUMMARY:
Objective: This study aimed to investigate the effect, onset and duration of action, and short-term outcomes of acupuncture therapy in the treatment of patients with severe chronic subjective tinnitus.

Methods: This study is a randomized, controlled trial evaluating patients with chronic, idiopathic and severe tinnitus. A total of 105 participants were divided into two groups using the randomization method: the study group that received real acupuncture therapy (n = 53) and the sham acupuncture group. Ten acupuncture sessions were applied over five weeks. After treatment, each participant was monitored for up to three months according to the changes in the Visual Analog Scale (VAS), Tinnitus Handicap Inventory (THI), Pure-Tone Audiometry and Speech Discrimination scores.

DETAILED DESCRIPTION:
This was a prospective, randomized, controlled study, approved by the local ethics committee and carried out in a single center in accordance with the ethical principles of the Helsinki Declaration (E-18-2165).

The inclusion criteria of the study for patients were determined as; (a) male and female patients aged 18 to 60 years, (b) unilateral or bilateral subjective tinnitus, (c) with a history of severe subjective tinnitus for at least one year, (d) patients with severe tinnitus according to the THI questionnaire result (over 38 points), (e) the patients who could not detect etiology of tinnitus in the otolaryngology examination, (f) not having received any treatment within the last six months. The patients who applied to the otorhinolaryngology clinic of our hospital were included in the study.

According to the randomization method, the group to which each participant was assigned was only known to the researcher who applied acupuncture therapy. The participants and the remaining researchers that administered THI to the participants were blinded to the groups.

The data were obtained from the patients' responses to VAS and THI questionnaires. Each participant completed the VAS and THI questionnaires seven times during the course of the five-week treatment and the three-month follow-up after treatment.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of the study for patients were determined as; (a) male and female patients aged 18 to 60 years, (b) unilateral or bilateral subjective tinnitus, (c) with a history of severe subjective tinnitus for at least one year, (d) patients with severe tinnitus according to the THI questionnaire result (over 38 points), (e) the patients who could not detect etiology of tinnitus in the otolaryngology examination, (f) not having received any treatment within the last six months. The patients who applied to the otorhinolaryngology clinic of our hospital were included in the study

Exclusion Criteria:

* The exclusion criteria were having received acupuncture therapy for the last three months for any reason, having a history of medication/surgery due to heart disease, having a disease that could cause objective tinnitus, such as Meniere's disease, otitis media, and otosclerosis, having metal allergy or needle phobia, having a history of psychotropic drug use, pregnancy or nursing, and not completing the THI survey.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-03-16 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
THI | 5 week
  tinnitus handicap index

SECONDARY OUTCOMES:
VAS | 5 week
  Visual Analog Scala

CONTACTS AND LOCATIONS:
Locations (1):
- Ihsan Kuzucu, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
A total of 179 subjects with chronic severe subjective tinnitus were initially evaluated. After applying the related criteria, 70 patients (39.1%) were excluded from the study. Of the remaining 109 participants (60.9%), 105 (92%) completed the study. The study group consisted of 53 participants, 19 male and 34 female, with a mean age of 50.70 ± 9.96 years. In the control group, there were 52 participants, 17 male and 35 female, with a mean age of 47.63 ± 11.35 years.

REFERENCES:
- See also: comparison acupuncture — https://www.ncbi.nlm.nih.gov/pubmed/29945669